CLINICAL TRIAL: NCT02352324
Title: Continuous Cardiac Output Monitoring Using esCCO: a Validation vs. Transpulmonary Thermodilution in Off-pump Coronary Artery Bypass Grafting
Brief Title: Cardiac Output Monitoring With Estimated Continuous Cardiac Output (esCCO) vs. Transpulmonary Thermodilution (TPTD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: esCCO-vs-TPTD
Record Dates: First submitted 2014-10-06; First posted 2015-02-02 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Pulse Wave Analysis
Keywords: cardiac output; coronary artery bypass grafting; minimally invasive hemodynamic monitoring; fluid responsiveness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluid responsiveness tests (Experimental): After the end of surgery in ICU the positive end-expiratory pressure (PEEP) test of 15 cm H2O for 300 seconds will be performed. Following PEEP test, the two-step fluid load test of 6 ml/kg balanced crystalloid solution will be performed sharing in two portions: Initial mini FLT (mFLT) of 1.5 ml/kg within 1 min (approximately 100 mL) followed by the registration of continuous CI and traditional fluid responsiveness parameters and the rest of standard FLT (4.5 mL/kg) within 5 minutes (approximately 350 mL) followed by transpulmonary thermodilution, registration of continuous cardiac index (CI) and classic fluid responsiveness parameters.
  Interventions: Other: Fluid responsiveness tests

INTERVENTIONS:
Other: Fluid responsiveness tests — After the end of surgery in ICU the positive end-expiratory pressure (PEEP) test of 15 cm H2O for 300 seconds will be performed. Following PEEP test, the two-step fluid load test of 6 ml/kg balanced crystalloid solution will be performed sharing in two portions: Initial mini FLT (mFLT) of 1.5 ml/kg within 1 min (approximately 100 mL) followed by the registration of continuous CI and traditional fluid responsiveness parameters and the rest of standard FLT (4.5 mL/kg) within 5 minutes (approximately 350 mL) followed by transpulmonary thermodilution, registration of continuous cardiac index (CI) and classic fluid responsiveness parameters.

SUMMARY:
The main goal of our study is to assess the accuracy and reproducibility of continuous beat-to-beat cardiac output (CO) measurement using pulse wave transit time in patients undergoing off-pump coronary artery bypass grafting.

DETAILED DESCRIPTION:
Using appropriate statistical methods the cardiac index values obtained via pulse wave transit time with esCCO system will be compared with traditional transpulmonary thermodilution technique.

ELIGIBILITY:
Inclusion Criteria:

* Elective isolated off-pump coronary arteries bypass grafting.
* Age > 18 years and < 80 yrs.
* Preoperative echocardiographic ejection fraction > 0.35

Exclusion Criteria:

* Simultaneous operation (carotid endarterectomy, ventricular aneurysm resection, etc.).
* Constant form of atrial fibrillation.
* Severe valve dysfunction.
* Peripheral vascular disease (including significant peripheral arteriopathy" which precludes the use of peripheral plethysmography).
* The surgical requirement to harvest both radial arteries.
* Intraaortic balloon pump.

Discontinuation Criteria:

* Transfer to cardiopulmonary bypass (on-pump CABG).
* The PEEP test will be discontinued before standard duration in patients with PEEP-induced profound MAP decrease below 50 mm Hg, bradycardia (< 50/min) or CIPCA < 1.9 l/min/m2 exceeding 1 minute.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Accuracy (between the method bias and angular bias) and precision (between the method standart deviation and radial limit of agreement) of esCCO cardiac output measurement | Up to 24 hrs post surgery
  Mean bias and standard deviation according to Bland-Altman analysis and angular bias and radial limit of agreement according to polar plot analysis for cardiac output assessed using pulse wave transit time in comparison with transpulmonary thermodilution

SECONDARY OUTCOMES:
Ability of augmented PEEP test (changes in cardiac output in response to an increase in PEEP) for predict the fluid responsiveness (changes in cardiac output in response to fluid load) in the early postoperative period | Immediate postoperatively
  Prediction of changes in cardiac output in response to fluid load in early postoperative period of off-pump CABG using the assessment of reaction of cardiac output to an increase in PEEP. Evaluation of correlation and ROC curve.
Ability of mini fluid load test (changes in CO in response to fast injection of minimal fluid volume) to predict fluid responsiveness (changes in CO in response to injection of standard fluid volume) in the immediate postoperative period following OPCAB | Immediate postoperatively
  Prediction of changes in cardiac output in response to fluid load in the immediate postoperative period following OPCAB using the assessment of reaction of cardiac output to an increase mini fluid load. Evaluation of correlation and ROC curve.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Y Kirov, MD, PhD, Study Director — Northern State Medical University; Alexey A Smetkin, MD, Principal Investigator — Northern State Medical University
Locations (1):
- Dep. of Anesthesiology, Northern SMU, Arkhangelsk, Russia